CLINICAL TRIAL: NCT00044174
Title: Dyadic Interactions in Depressed and Non-Depressed Mothers With Their Infants
Brief Title: Dyadic Interactions in Depressed and Non-Depressed Mothers and Their Infants
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020278; 02-CH-0278
Record Dates: First submitted 2002-08-20; First posted 2002-08-21 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12-19

CONDITIONS: Depression
Keywords: Infant; maternal health; Natural History
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Depressed Mothers/Infants: Mothers and their 5 month old infants who have been clinically diagnosed as exhibiting depressive symptoms
- Non-depressed Mothers/Infants: Mothers and their 5 month old infants who have been clinically diagnosed as not exhibiting depressive symptoms

SUMMARY:
This study will examine 1) differences among mothers behaviors and how these behaviors influence their infants reactions, and 2) how mother-child interactions relate to children s temperament, and cognitive (thought processing) abilities, and other areas of development.

Depressed and non-depressed English-speaking mothers between 20 and 45 years of age, with an infant 4 months or younger, may be eligible for this study. Candidates will be screened with a mailed survey regarding their moods and feelings. Participants will undergo the following procedures:

* Psychiatric Interview: Subjects will participate in a 30-90 minute interview consisting of a series of standardized questions about the their behaviors and feelings. Participants whose interviews suggest a condition that may impact their mental health will be referred to the study clinician for follow-up to confirm or clarify the preliminary findings. Continued participation in the study will be determined following this.
* Home Visit: A study investigator will visit the home for 1 hour to film the mother and baby during the mother s typical daily activities. This visit will take place when the baby is about 5 months old. At the end of the visit, the mother will be given a variety of surveys to fill out at home and return at the next visit (see Lab Visit below). The survey questions deal with the mother s relationship with her partner, support from people in her life, typical behaviors of her infant, and how often she feels certain emotions. A packet of surveys will also be left for the participant s partner to complete and mail back to the investigator. The partner may or may not be the child s biological father and may or may not choose to participate in the study.
* Lab Visit: Within 1 week of the home visit, the mother and child will come to the NICHD clinic for about 2 hours. During this time, the mother will return the previous surveys and fill out another one regarding her current mood. She will then interact with her child, who will be seated in front of her. The 20-minute session will be videotaped. (There will be breaks during the session.) The mother will be instructed about how she should act (happy or sad). She and her baby will then participate in a variety of filmed situations that will induce certain emotions in the baby, such as happiness, fear, activity, frustration, and interest, in order to learn how different children react to different situations.

Participants will be contacted to continue the study when their babies are 12 months old and again when the children are 24 months old. The above procedures will be repeated and some new measures will be added for toddlers that involve activities investigating aspects of early language and social reasoning..

DETAILED DESCRIPTION:
Maternal depression is a concurrent and longitudinal risk factor for children s development. Maternal depression exerts direct effects and indirect effects through proximal processes of mother-child dyadic interactions. Both depressed mothers and their infants are inattentive, unresponsive, affectively flat, and disengaged during naturalistic interactions, and their dyadic interactions have been described as less synchronous. Our primary objective is to investigate differences between depressed and non-depressed dyads in maternal behaviors, child behaviors, and dyadic behaviors in terms of latency, synchrony, and contingency. In the present study, we propose to examine the determinants and effects of dyadic interactions of depressed and nondepressed mothers with their infants across several domains of child development. We plan to replicate and extend previous work by observing the dyads in naturalistic as well as experimental face-to-face settings at 5, 12, and 24 months.

Groups of depressed and nondepressed mothers will be selected on the basis of self-reports of depressive symptoms and by clinical diagnostic interviews. These assessments will be repeated at 12 and 24 months to assess the course of maternal depression. The study consists of a home visit, a lab visit, and administration of questionnaires to mothers and their spouses or partners at three time points. All maternal and child behaviors during dyadic interactions will be coded as continuous streams of data for analysis of reciprocal influences within the dyad. By coding a range of behaviors such as facial affect, vocalization, physical activity, and visual attention of the mother and infant, we hope to capture variations in mother-child interactions, both between and within depressed and nondepressed dyads. Differences in styles of dyadic interactions have been shown to have important consequences on subsequent child development in several domains. In addition, experimental simulations will consist of instructed 'depressed' and 'happy' simulations of mothers with their infants. Specific simulations allow observation of changes in infant behaviors from the spontaneous episodes and comparison between depressed and nondepressed dyads.

Understanding the context of child development, both normative and atypical, is important as means of elucidating the processes by which maternal depression operates as a risk factor for children s cognitive and socioemotional development. Several socio-demographic and psychosocial factors will be assessed by maternal and paternal self-reports to examine which factors exacerbate or buffer the effects of maternal depression. In addition to modifying the observations of maternal and child behaviors to be age-appropriate, new measures will be introduced at 12 and 24 months to capture child s functioning in multiple areas.

ELIGIBILITY:
* INCLUSION CRITERIA:

Mothers and infants must meet certain criteria to be included in the study. Selection criteria are: maternal age between 20 and 45 years, ability to read and write in English, normal pregnancy/delivery status without birth complications, term birth (+/- 14 days from due date), and singleton status of the child. Approximately equal numbers of male and female infants will be recruited, and to the extent possible, the two groups of depressed and nondepressed mothers will be matched on ethnic composition. Participants will be seen at 5, 12, and 24 months.

EXCLUSION CRITERIA:

None

Min Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Depressed and non-depressed English-speaking mothers between 20 and 45 years of age, with an infant 4 months or younger, may be eligible for this study. Candidates will be screened with a mailed survey regarding their moods and feelings.
Sampling Method: Non-Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2002-08-20 (Actual)

PRIMARY OUTCOMES:
Multiple measures of child cognitive and socioemotional development as well as maternal psychosocial factors | When child is 5, 12, and 24 months
  Our primary objective is to investigate differences between depressed and non-depressed dyads in maternal behaviors, child behaviors, and dyadic behaviors in terms of latency, synchrony, and contingency. In the present study, we propose to examine the determinants and effects of dyadic interactions of depressed and nondepressed mothers with their infants across several domains of child development. We plan to replicate and extend previous work by observing the dyads in naturalistic as well as experimental face-to-face settings at 5, 12, and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Putnick, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-CH-0278.html